CLINICAL TRIAL: NCT06242405
Title: Efficacy and Safety of Different Frequencies of Human Umbilical Cord-mesenchymal Stem Cells Through Peripheral Vein in Patients with End-stage Liver Disease
Brief Title: Effect of Different Frequencies of Umbilical Cord-mesenchymal Stem Cells Through Peripheral Vein in Patients with ESLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHNKKY-DFSC
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: End-Stage Liver DIsease
Keywords: cirrhosis; end-stage liver diseases; umbilical cord-mesenchymal stem cells; randomized controlled trial
MeSH Terms: conditions — End Stage Liver Disease; Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-infusion group (Experimental): Single peripheral venous infusion of stem cells
  Interventions: Biological: umbilical cord-mesenchymal stem cells
- Double-infusion group (Experimental): Repeated peripheral venous infusion of stem cells within one month
  Interventions: Biological: umbilical cord-mesenchymal stem cells

INTERVENTIONS:
Biological: umbilical cord-mesenchymal stem cells — Umbilical cord mesenchymal stem cells injected through peripheral veins
  Other Names: UC-MSCs

SUMMARY:
Stem cells are non-terminal cells that can self renew and replicate through symmetric or asymmetric division, with the potential to differentiate into different types of cells and tissues. Multiple studies have shown that mesenchymal stem cell has good safety and effectiveness in improving acute or chronic liver injury. Randomized controlled trials have confirmed the efficacy of single infusion of stem cells in treating ESLD. It seems that the multiple infusion is better than single infusion.

DETAILED DESCRIPTION:
Ninety-two participants with end-stage liver disease admitted to the Department of Gastroenterology of the General Hospital of Northern Theater Command are expected to be enrolled over a period of 1 year. The participants will be randomly divided into single-infusion and double-infusion stem cell groups by peripheral vein. The investigators will observe alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, albumin, prothrombin time, international normalized ratio, model for end-stage liver disease score, and Child-Pugh score in patients at weeks 24 post-infusion.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-80 years old
* 2. End-stage liver disease
* 3. Signed informed consent

Exclusion Criteria:

* 1. Tumours of the liver or other organs
* 2. Liver transplantation recipients
* 3. Acute myocardial infarction, acute heart failure, type I and type II respiratory failure, pulmonary embolism, acute cerebral infarction, acute cerebral haemorrhage and other serious cardiopulmonary diseases
* 4. Other diseases that may seriously affect the survival
* 5. Human immunodeficiency syndrome
* 6. Interferon or glucocorticoid therapy within 1 year
* 7. Treated for mental illness
* 8. Participation in other clinical trials within 30 days
* 9. Pregnant or breastfeeding subjects
* 10. Allergic asthma, allergic urticaria, eczema, or a history of multiple drug and food allergies
* 11. Other circumstances that are unsuitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Child A | 24 weeks
  Patients with Child A

SECONDARY OUTCOMES:
Change in liver function parameters | 24 weeks
  Values of alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, serum albumin, prothrombin time, and international normalized ratio and the scores of MELD and Child-Pugh
Incidence of hepatic decompensation events | 24 weeks
  Number of patients who will develop gastrointestinal bleeding, ascites and hepatic encephalopathy
Survival rate and liver transplant rate | 24 weeks
  Number of patients surviving and undergoing liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, MD, Study Director — The General Hospital of Northern Theater Command; Wen Ning, MM, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volarevic V, Nurkovic J, Arsenijevic N, Stojkovic M. Concise review: Therapeutic potential of mesenchymal stem cells for the treatment of acute liver failure and cirrhosis. Stem Cells. 2014 Nov;32(11):2818-23. doi: 10.1002/stem.1818. PMID 25154380
- [Background] Wang J, Li Q, Li W, Mendez-Sanchez N, Liu X, Qi X. Stem Cell Therapy for Liver Diseases: Current Perspectives. Front Biosci (Landmark Ed). 2023 Dec 28;28(12):359. doi: 10.31083/j.fbl2812359. PMID 38179765